CLINICAL TRIAL: NCT07122050
Title: Safety and Effectiveness of Prizvalve Transcatheter Aortic Valve in Patients With Failing Bioprosthetic Valves
Brief Title: Prizvalve Transcatheter Aortic Valve in Failing Bioprosthetic Valves
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prizvalve-VIV-202504
Record Dates: First submitted 2025-07-22; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Failing Bioprosthetic Valves
Keywords: Prizvalve Valve in Valve

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 105 Failing Mitral Bioprosthetic Valve (Experimental)
  Interventions: Device: Prizvalve® system Transcatheter valve-in-valve replacement
- At Least 10 Failing Tricuspid Bioprosthetic Valve (Experimental)
  Interventions: Device: Prizvalve® system Transcatheter valve-in-valve replacement
- At Least 10 Failing Aortic Bioprosthetic Valve (Experimental)
  Interventions: Device: Prizvalve® system Transcatheter valve-in-valve replacement

INTERVENTIONS:
Device: Prizvalve® system Transcatheter valve-in-valve replacement — Transcatheter valve-in-valve replacement procedure was performed according to standard clinical practice. Successful vascular access, delivery and deployment of the device and successful retrieval of the delivery system will be attempted.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the Prizvalve transcatheter aortic valve in subjects who are at high or greater risk with failing bioprosthetic valves.

DETAILED DESCRIPTION:
Prospective, single arm, multicenter study

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation:

1. Age≥18 years old;
2. Failing bioprosthetic valve (≥moderate stenosis and/or ≥moderate regurgitation);
3. NYHA Function Class≥ II;
4. Patient who is anatomically suitable for the implantation of the Prizvalve®;
5. According to heart team , patient is at high or greater surgical risk or not suitable for redo open heart surgery of valve replacement;
6. Patient understands the purpose of the trial and volunteers to participate in, sign the informed consent form and is willing to accept relevant examinations and clinical follow-ups.

Exclusion Criteria:

1. Moderate or greater paravalvular regurgitation of the degenerated bioprosthetic valve；
2. Degenerated valve that cannot be securely fixed within the native annulus or exhibits structural incompleteness；
3. Anatomical features deemed unsuitable for transcatheter implantation.
4. Anatomical features that significantly increase the risk of left ventricular outflow tract (LVOT) obstruction；
5. Acute myocardial infarction within 30 days prior to enrollment；
6. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation；
7. Active infective endocarditis or any other active infection；
8. Severe right ventricular dysfunction or severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20 %；
9. Inability to tolerate anticoagulant or antiplatelet therapy；
10. Cerebrovascular accident within 3 months prior to enrollment, excluding transient ischemic attack；
11. Refusal to undergo emergency cardiac surgery under any circumstances；
12. Participation in another drug or device clinical trial that has not yet reached its primary endpoint as of the time of enrollment；
13. Investigator-assessed poor compliance that would preclude adherence to protocol requirements；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | At 30 days
  The primary end point is the 30 days all-cause mortality

SECONDARY OUTCOMES:
Device success | immediate post-surgical
  Device Success Criteria
  1. Successful vascular access, delivery, deployment and implantation of the study device, with complete removal of the delivery system from the body;
  2. The implanted prosthetic valve achieves the intended haemodynamic performance, defined as the absence of moderate or greater prosthetic valve stenosis or regurgitation.
Procedural success | immediate post-surgical
  Procedural Success Criteria
  1. Correct anatomical positioning of the implanted valve;
  2. No intra-operative or immediate post-procedural death (≤ 72 h);
  3. Achievement of the intended therapeutic goal without occurrence of any major intra-operative complication, including but not limited to coronary obstruction, ventricular septal perforation, damage or dysfunction of other native valves, cardiac tamponade, procedure termination, or conversion to open cardiac surgery.
All-cause mortality | At 6 months, 1 year
The incidence of rehospitalization | At 30 days, 6 months, 1 year
The incidence of myocardial infarction | At 30 days, 6 months, 1 year
The incidence of stroke | At 30 days, 6 months, 1 year
The incidence of bleeding | At 30 days, 6 months, 1 year
The incidence of acute kidney injury | At 30 days, 6 months, 1 year
The incidence of permanent pacemaker implantation | At 30 days, 6 months, 1 year
The incidence of vascular and access-related complications | At 30 days, 6 months, 1 year
The incidence of procedure-related complications | At 30 days, 6 months, 1 year
The incidence of valve dysfunction | At 30 days, 6 months, 1 year
The incidence of NYHA functional class improvement | At 30 days, 6 months, 1 year
  the New York Heart Association to quantify the severity of functional limitation and symptoms attributable to cardiac disease
The incidence of quality-of-life improvement | At 30 days, 6 months, 1 year
  By SF-12 Health Survey (Short-Form 12-item Health Survey)
The incidence of major adverse cardiovascular and cerebrovascular events (MACCE) | At 30 days, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yang, MD, PhD, Principal Investigator — Department of Cardiovascular Surgery of Xijing Hospital, Air Force Military Medical University
Locations (1):
- Department of Cardiovascular Surgery of Xijing Hospital, Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) would not be shared, according to local authority data privacy policy.